CLINICAL TRIAL: NCT01318473
Title: A Prospective, Open-Label, Single-Arm, Single-Center Study Evaluating the Use of the ActiSight™ Needle Guidance System in Patients Undergoing CT-Guided Percutaneous Chest Aspiration and Biopsy With Lesions Smaller Than 15 mm
Brief Title: The Use of the ActiSight™ Needle Guidance System in Patients Undergoing CT-Guided With Lesions Smaller Than 15 mm
Acronym: ActiSight
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASNG-LFNA-102-IL; ASNG-LFNA-101-IL (Other: Protocol #)
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ActiSight™ Needle Guidance System (Other): ActiSight™ Needle Guidance System is comprised of several sub-system components: a computer, a disposable ActiSensor optical sensor, and the disposable ActiSticker, which provides a reference for the insertion of the tool and for the camera.
  Interventions: Device: ActiSight™ Needle Guidance System

INTERVENTIONS:
Device: ActiSight™ Needle Guidance System — ActiSight™ Needle Guidance System is comprised of several sub-system components: a computer, a disposable ActiSensor optical sensor, and the disposable ActiSticker, which provides a reference for the insertion of the tool and for the camera.
  Other Names: ActiSight System

SUMMARY:
This will be a prospective, single-arm, single-center, open-label study to evaluate the use of the ActiSight™ Needle Guidance System in patients with lung lesions smaller than 15 mm undergoing CT-guided percutaneous chest aspiration.

Target location will be in the chest area; the procedure will be performed by a trained physician.

DETAILED DESCRIPTION:
Subjects who are scheduled for clinically indicated percutaneous chest aspiration/biopsy procedures will be screened for inclusion in the study.

Within an 18-day screening period, eligible subjects will be enrolled into the study and undergo percutaneous chest aspiration or percutaneous biopsy utilizing the ActiSight™ Needle Guidance system using CT to guide the needle. Subjects will be followed-up for at least one hour at the clinic for safety and preliminary accuracy evaluations. An erect chest radiograph will be performed within 90 minutes of observation after the chest aspiration to detect the majority of post procedure pneumothoraces. A follow-up visit will be conducted within 7-10 days after the procedure day for safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older at the time of enrollment
* Subjects scheduled for clinically indicated percutaneous chest aspiration/biopsy procedures
* Subjects with lung lesions less than 15 mm.
* Written informed consent to participate in the study
* Ability to comply with the requirements of the study procedures

Exclusion Criteria:

* Subjects who cannot tolerate mild sedation
* Subjects who participated in an active stage of any drug, intervention or treatment trial within 30 days of enrollment.
* Subjects with preexisting conditions which, in the opinion of the investigator, interfere with the conduct of the study.
* Subjects who are uncooperative or cannot follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Frequency of adequate sample for diagnosis obtained in the procedure as determined from the Histology / Cytology report | 6 month
  Frequency of adequate sample for diagnosis obtained in the procedure as determined from the Histology / Cytology report

SECONDARY OUTCOMES:
Frequency of target reached by the biopsy or aspiration tool, as determined by a qualified physician reviewing the CT images | 6 month
  Frequency of target reached by the biopsy or aspiration tool, as determined by a qualified physician reviewing the CT images
Number of needle punctures through the skin | 6 month
  Number of needle punctures through the skin
Number of needle punctures through the pleura | 6 month
  Number of needle punctures through the pleura
Number of CT scans needed | 6 month
  Number of CT scans needed
Duration of procedure: patient preparation, planning, guidance and Cytolog report. | 6 month
  Duration of procedure: patient preparation, planning, guidance and Cytolog report.

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Tiran, Dr., Principal Investigator — Tel-Aviv Sourasky Medical Center